CLINICAL TRIAL: NCT07220135
Title: A Randomized Trial of Neoadjuvant THP vs TCHP for HER2-amplified/Positive Breast Cancer (NeoTHERa)
Brief Title: Trial of Neoadjuvant THP vs TCHP for HER2-Amplified/Positive Breast Cancer
Acronym: NeoTHERa
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Yiduo Hu, MD, PhD, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2025-NeoTHERa
Record Dates: First submitted 2025-10-13; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Docetaxel; Trastuzumab; Biosimilar Pharmaceuticals; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Other): Carboplatin and docetaxel plus trastuzumab and pertuzumab every 21 days for 6 cycles. Doses and route of administration per institutional standards.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Drug: Trastuzumab (or biosimilar); Drug: Pertuzumab (or biosimilar)
- Arm B (Other): Docetaxel plus trastuzumab and pertuzumab every 21 days for 6 cycles. Doses and route of administration per institutional standards.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab (or biosimilar); Drug: Pertuzumab (or biosimilar)

INTERVENTIONS:
Drug: Carboplatin — All of the treatment being received by the study participants during the course of the study is standard of care.
  Other Names: Paraplatin
  Arms: Arm A
Drug: Docetaxel — All of the treatment being received by the study participants during the course of the study is standard of care.
  Other Names: Taxotere
Drug: Trastuzumab (or biosimilar) — All of the treatment being received by the study participants during the course of the study is standard of care.
  Other Names: Herceptin
Drug: Pertuzumab (or biosimilar) — All of the treatment being received by the study participants during the course of the study is standard of care.
  Other Names: Perjeta

SUMMARY:
This is a randomized phase II study to evaluate the pathological complete response (pCR) rate with two neoadjuvant regimens (Docetaxel+Carboplatin+Herceptin/Perjeta and Docetaxel+Herceptin/Perjeta) in HER2 amplified/positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* 18 years of age or older
* Histologically confirmed cT2-T3 N0-N2, cT1 N1-N2, or cTX N1-N2 HER2 positive breast cancer (The invasive tumor must be HER2-positive based on the current ASCO-CAP guidelines; Patients are eligible regardless of estrogen receptor (ER) or progesterone receptor (PR) expression status. However, percentage of both ER and PR positivity must be documented in the pathology report.)
* No previous ipsilateral breast surgery for the current breast cancer
* No previous chemotherapy, anti-HER2 therapy, immunotherapy, endocrine therapy, or radiotherapy for the current breast cancer
* ECOG Performance Status 0-1 documented within 28 days prior to the start of study treatment (Appendix A)
* Breast and axillary imaging (including mammogram, ultrasound and/or MRI, per standard of care) within 49 days (7 weeks) prior to treatment initiation
* Subjects with clinically and/or radiographically abnormal axillary or internal mammary lymph nodes should have pathologic confirmation of disease status with image-guided biopsy or fine needle aspiration unless deemed medically unsafe
* Co-enrollment in the PRO-HER2 (HSC #160944) observational registry protocol
* Archival breast tumor tissue has been obtained or has been requested for use, which should include either a formalin-fixed paraffin-embedded (FFPE) block, or sixteen slides (fourteen 5-micron uncharged unstained slides plus either two H&E slides or two 5-micron charged unstained slides) - from primary breast tumor only.
* Subjects with bilateral synchronous HER2 positive breast cancer are eligible if they meet other eligibility criteria
* Neuropathy: No baseline grade 2 or above neuropathy
* Not pregnant, not breastfeeding, and at least one of the following applies: Not a woman of reproductive potential as defined by institutional standards; A woman of reproductive potential who agrees to follow contraceptive guidelines per institutional standards
* Adequate organ function, defined as follows: Hematologic (assessed ≤ 21 days of treatment initiation): Absolute neutrophil count ≥ 1,500/μL (with the exception of patients with documented Fy(a-/b-) (Duffy null) immunophenotype, in which case absolute neutrophil count ≥1,200/uL is allowed), Platelets ≥ 100,000/μL, Leukocytes ≥ 3,000/μL, Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (must be met without erythropoietin dependency and without erythrocyte transfusion within the last two weeks); Hepatic (assessed ≤ 21 days of treatment initiation): Total bilirubin ≤ 1.5x ULN, AST(SGOT) and ALT(SPGT) ≤ 2x ULN, Serum albumin ≥ 3.0 g/dL; Cardiac (assessed ≤ 49 days of treatment initiation): Normal baseline echocardiogram or MUGA scan including LVEF ≥ 50%, per standard of care

Exclusion Criteria:

* Current or anticipated use of other investigational agents while participating in this study
* Clinically or radiographically detected metastatic disease
* Inflammatory breast cancer
* Prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the treatment regimen. Note: Patients with squamous cell or basal cell carcinoma of the skin, ductal carcinoma in situ (DCIS) of the breast, or carcinoma in situ (CIS) of the uterine cervix who have undergone definitive therapy are not excluded from participation
* History of allergic reactions attributed to carboplatin, docetaxel, trastuzumab, or pertuzumab
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of this study, interfere with the subject's participation for the full duration of the study, or it is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Pregnancy, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. There is a potential for congenital abnormalities and for this regimen to harm breastfeeding infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-14 (Estimated); Primary Completion 2027-11-14 (Estimated); Study Completion 2031-05-14 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate in the breast and axilla in the two treatment arms | At time of breast surgery
  To evaluate the pathological complete response (pCR) rate with two neoadjuvant regimens (Docetaxel+Carboplatin+Herceptin+Perjeta (TCHP) and Docetaxel+Herceptin+Perjeta (THP)) in HER2+ breast cancer.

SECONDARY OUTCOMES:
Residual cancer burden (RCB) | At time of breast surgery
  Determine residual cancer burden (RCB) 0+1 rate
Assess the toxicity and tolerability of each regimen | Start of study treatment (6 cycles every 21 days) until 30 days after last dose of study treatment.
  Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0. Only grade 3 and higher CTCAE toxicities will be collected. Alopecia of any grade will not be collected.
HER2DX pathological complete response (pCR) score status | Results of HER2DX testing are expected to be available within 3-6 weeks of submission of FFPE samples
  Assess pathological complete response (pCR) and residual cancer burden (RCB) by HER2DX pCR score status. The HER2DX test reports three pCR Likelihood Groups for response (High, Medium and Low).
Recurrence-Free Survival (RFS) | From 3- and 5-years from diagnosis
  RFS is defined as the time from diagnosis to first recurrence (invasive ipsilateral breast, invasive local/regional, or distant), or to death as a result of any cause.
Event-Free Survival (EFS) | From 3- and 5-years from diagnosis
  EFS is defined as the time from diagnosis to first recurrence (invasive ipsilateral breast, invasive local/regional, or distant) or to breast cancer-related death.
Overall Survival (OS) | From 3- and 5-years from diagnosis
  OS is defined as the time from diagnosis to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yiduo Hu, MD, Principal Investigator — University of Kansas Medical Center

REFERENCES:
- [Background] Harris, J., M. Morrow, and L. Norton, Malignant tumors of the breast, in Cancer: principles and practice of oncology, V.J. DeVita, S. Hellman, and S. Rosenberg, Editors. 1997, Lippincott-Raven: Philadelphia. p. 1557-1602.
- [Background] Untch M, Rezai M, Loibl S, Fasching PA, Huober J, Tesch H, Bauerfeind I, Hilfrich J, Eidtmann H, Gerber B, Hanusch C, Kuhn T, du Bois A, Blohmer JU, Thomssen C, Dan Costa S, Jackisch C, Kaufmann M, Mehta K, von Minckwitz G. Neoadjuvant treatment with trastuzumab in HER2-positive breast cancer: results from the GeparQuattro study. J Clin Oncol. 2010 Apr 20;28(12):2024-31. doi: 10.1200/JCO.2009.23.8451. Epub 2010 Mar 22. PMID 20308670
- [Background] Broglio KR, Quintana M, Foster M, Olinger M, McGlothlin A, Berry SM, Boileau JF, Brezden-Masley C, Chia S, Dent S, Gelmon K, Paterson A, Rayson D, Berry DA. Association of Pathologic Complete Response to Neoadjuvant Therapy in HER2-Positive Breast Cancer With Long-Term Outcomes: A Meta-Analysis. JAMA Oncol. 2016 Jun 1;2(6):751-60. doi: 10.1001/jamaoncol.2015.6113. PMID 26914222
- [Background] Bear HD. Indications for neoadjuvant chemotherapy for breast cancer. Semin Oncol. 1998 Apr;25(2 Suppl 3):3-12. No abstract available. PMID 9566201
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 1998 Aug;16(8):2672-85. doi: 10.1200/JCO.1998.16.8.2672. PMID 9704717
- [Background] Kuerer HM, Newman LA, Smith TL, Ames FC, Hunt KK, Dhingra K, Theriault RL, Singh G, Binkley SM, Sneige N, Buchholz TA, Ross MI, McNeese MD, Buzdar AU, Hortobagyi GN, Singletary SE. Clinical course of breast cancer patients with complete pathologic primary tumor and axillary lymph node response to doxorubicin-based neoadjuvant chemotherapy. J Clin Oncol. 1999 Feb;17(2):460-9. doi: 10.1200/JCO.1999.17.2.460. PMID 10080586
- [Background] Green M, Hortobagyi GN. Neoadjuvant chemotherapy for operable breast cancer. Oncology (Williston Park). 2002 Jul;16(7):871-84, 889; discussion 889-90, 892-4, 897-8. PMID 12164555
- [Background] van der Hage JA, van de Velde CJ, Julien JP, Tubiana-Hulin M, Vandervelden C, Duchateau L. Preoperative chemotherapy in primary operable breast cancer: results from the European Organization for Research and Treatment of Cancer trial 10902. J Clin Oncol. 2001 Nov 15;19(22):4224-37. doi: 10.1200/JCO.2001.19.22.4224. PMID 11709566
- [Background] Valero V, Buzdar AU, McNeese M, Singletary E, Hortobagyi GN. Primary chemotherapy in the treatment of breast cancer: the University of Texas M. D. Anderson Cancer Center experience. Clin Breast Cancer. 2002 Oct;3 Suppl 2:S63-8. doi: 10.3816/cbc.2002.s.014. PMID 12435294
- [Background] Wang J, Buchholz TA, Middleton LP, Allred DC, Tucker SL, Kuerer HM, Esteva FJ, Hortobagyi GN, Sahin AA. Assessment of histologic features and expression of biomarkers in predicting pathologic response to anthracycline-based neoadjuvant chemotherapy in patients with breast carcinoma. Cancer. 2002 Jun 15;94(12):3107-14. doi: 10.1002/cncr.10585. PMID 12115341
- [Background] Cortazar, P., et al., Meta-analysis results from the collaborative trials in neoadjuvant breast cancer (CTNeoBC) [abstract]. Cancer Res, 2012. 72(24 Suppl): p. Abstract nr P1-14-20.
- [Background] Slamon D, Eiermann W, Robert N, Pienkowski T, Martin M, Press M, Mackey J, Glaspy J, Chan A, Pawlicki M, Pinter T, Valero V, Liu MC, Sauter G, von Minckwitz G, Visco F, Bee V, Buyse M, Bendahmane B, Tabah-Fisch I, Lindsay MA, Riva A, Crown J; Breast Cancer International Research Group. Adjuvant trastuzumab in HER2-positive breast cancer. N Engl J Med. 2011 Oct 6;365(14):1273-83. doi: 10.1056/NEJMoa0910383. PMID 21991949
- [Background] Schneeweiss A, Chia S, Hickish T, Harvey V, Eniu A, Hegg R, Tausch C, Seo JH, Tsai YF, Ratnayake J, McNally V, Ross G, Cortes J. Pertuzumab plus trastuzumab in combination with standard neoadjuvant anthracycline-containing and anthracycline-free chemotherapy regimens in patients with HER2-positive early breast cancer: a randomized phase II cardiac safety study (TRYPHAENA). Ann Oncol. 2013 Sep;24(9):2278-84. doi: 10.1093/annonc/mdt182. Epub 2013 May 22. PMID 23704196
- [Background] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Background] Villacampa G, Matikas A, Oliveira M, Prat A, Pascual T, Papakonstantinou A. Landscape of neoadjuvant therapy in HER2-positive breast cancer: a systematic review and network meta-analysis. Eur J Cancer. 2023 Sep;190:112885. doi: 10.1016/j.ejca.2023.03.042. Epub 2023 Apr 8. PMID 37142539
- [Background] Lin B, Fan J, Liu F, Wen Y, Li J, Gao F, Zhang Y, Feng G, Du X, Chen W. Efficacy and Safety of Dual Anti-HER2 Blockade and Docetaxel With or Without Carboplatin as Neoadjuvant Regimen for Treatment of HER2-Positive Breast Cancer. Technol Cancer Res Treat. 2023 Jan-Dec;22:15330338231218152. doi: 10.1177/15330338231218152. PMID 38031361
- [Background] Lv M, Guo H, Wang C, Tian P, Ma Y, Chen X, Luo S. Neoadjuvant docetaxel with or without carboplatin plus dual HER2 blockade for HER2-positive breast cancer: a retrospective multi-center Chinese study. Gland Surg. 2020 Dec;9(6):2079-2090. doi: 10.21037/gs-20-791. PMID 33447559
- [Background] Waks AG, Desai NV, Li T, Poorvu PD, Partridge AH, Sinclair N, Spring LM, Faggen M, Constantine M, Metzger O, Alberti J, Deane J, Rosenberg SM, Frank E, Tolaney SM, Krop IE, Tung NM, Tayob N, King TA, Mittendorf EA, Winer EP. A prospective trial of treatment de-escalation following neoadjuvant paclitaxel/trastuzumab/pertuzumab in HER2-positive breast cancer. NPJ Breast Cancer. 2022 May 10;8(1):63. doi: 10.1038/s41523-022-00429-7. PMID 35538105
- [Background] Chen XC, Jiao DC, Qiao JH, Wang CZ, Sun XF, Lu ZD, Li LF, Zhang CJ, Yan M, Wei Y, Chen B, Feng YQ, Deng M, Ma MD, Plichta JK, He YW, Liu ZZ. De-escalated neoadjuvant weekly nab-paclitaxel with trastuzumab and pertuzumab versus docetaxel, carboplatin, trastuzumab, and pertuzumab in patients with HER2-positive early breast cancer (HELEN-006): a multicentre, randomised, phase 3 trial. Lancet Oncol. 2025 Jan;26(1):27-36. doi: 10.1016/S1470-2045(24)00581-3. Epub 2024 Nov 26. PMID 39612919
- [Background] Gianni L, Pienkowski T, Im YH, Roman L, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi G, Szado T, Ratnayake J, Ross G, Valagussa P. Efficacy and safety of neoadjuvant pertuzumab and trastuzumab in women with locally advanced, inflammatory, or early HER2-positive breast cancer (NeoSphere): a randomised multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Jan;13(1):25-32. doi: 10.1016/S1470-2045(11)70336-9. Epub 2011 Dec 6. PMID 22153890
- [Background] Ismael G, Hegg R, Muehlbauer S, Heinzmann D, Lum B, Kim SB, Pienkowski T, Lichinitser M, Semiglazov V, Melichar B, Jackisch C. Subcutaneous versus intravenous administration of (neo)adjuvant trastuzumab in patients with HER2-positive, clinical stage I-III breast cancer (HannaH study): a phase 3, open-label, multicentre, randomised trial. Lancet Oncol. 2012 Sep;13(9):869-78. doi: 10.1016/S1470-2045(12)70329-7. Epub 2012 Aug 9. PMID 22884505
- [Background] Tan AR, Im SA, Mattar A, Colomer R, Stroyakovskii D, Nowecki Z, De Laurentiis M, Pierga JY, Jung KH, Schem C, Hogea A, Badovinac Crnjevic T, Heeson S, Shivhare M, Kirschbrown WP, Restuccia E, Jackisch C; FeDeriCa study group. Fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection plus chemotherapy in HER2-positive early breast cancer (FeDeriCa): a randomised, open-label, multicentre, non-inferiority, phase 3 study. Lancet Oncol. 2021 Jan;22(1):85-97. doi: 10.1016/S1470-2045(20)30536-2. Epub 2020 Dec 21. PMID 33357420
- [Background] Bueno-Muino C, Echavarria I, Lopez-Tarruella S, Roche-Molina M, Del Monte-Millan M, Massarrah T, Jerez Y, Ayala de la Pena F, Garcia-Saenz JA, Moreno F, Rodriguez-Lescure A, Malon-Gimenez D, Ballesteros Garcia AI, Marin-Aguilera M, Galvan P, Braso-Maristany F, Waks AG, Tolaney SM, Mittendorf EA, Vivancos A, Villagrasa P, Parker JS, Perou CM, Pare L, Villacampa G, Prat A, Martin M. Assessment of a Genomic Assay in Patients With ERBB2-Positive Breast Cancer Following Neoadjuvant Trastuzumab-Based Chemotherapy With or Without Pertuzumab. JAMA Oncol. 2023 Jun 1;9(6):841-846. doi: 10.1001/jamaoncol.2023.0187. PMID 37103916
- [Background] Villacampa G, Tung NM, Pernas S, Pare L, Bueno-Muino C, Echavarria I, Lopez-Tarruella S, Roche-Molina M, Del Monte-Millan M, Marin-Aguilera M, Braso-Maristany F, Waks AG, Pascual T, Martinez-Saez O, Vivancos A, Conte PF, Guarneri V, Vittoria Dieci M, Griguolo G, Cortes J, Llombart-Cussac A, Munoz M, Vidal M, Adamo B, Wolff AC, DeMichele A, Villagrasa P, Parker JS, Perou CM, Fernandez-Martinez A, Carey LA, Mittendorf EA, Martin M, Prat A, Tolaney SM. Association of HER2DX with pathological complete response and survival outcomes in HER2-positive breast cancer. Ann Oncol. 2023 Sep;34(9):783-795. doi: 10.1016/j.annonc.2023.05.012. Epub 2023 Jun 9. PMID 37302750
- [Background] Llombart-Cussac A, Perez-Garcia J, Braso-Maristany F, Pare L, Villacampa G, Gion M, Schmid P, Colleoni M, Borrego MR, Galvan P, Parker JS, Buckingham W, Perou CM, Villagrasa P, Guerrero JA, Sampayo-Cordero M, Mancino M, Prat A, Cortes J. HER2DX Genomic Assay in HER2-Positive Early Breast Cancer Treated with Trastuzumab and Pertuzumab: A Correlative Analysis from the PHERGain Phase II Trial. Clin Cancer Res. 2024 Sep 13;30(18):4123-4130. doi: 10.1158/1078-0432.CCR-24-0464. PMID 38995291
- [Background] Waks AG, Ogayo ER, Pare L, Marin-Aguilera M, Braso-Maristany F, Galvan P, Castillo O, Martinez-Saez O, Vivancos A, Villagrasa P, Villacampa G, Tarantino P, Desai N, Guerriero J, Metzger O, Tung NM, Krop IE, Parker JS, Perou CM, Prat A, Winer EP, Tolaney SM, Mittendorf EA. Assessment of the HER2DX Assay in Patients With ERBB2-Positive Breast Cancer Treated With Neoadjuvant Paclitaxel, Trastuzumab, and Pertuzumab. JAMA Oncol. 2023 Jun 1;9(6):835-840. doi: 10.1001/jamaoncol.2023.0181. PMID 37103927
- [Background] Yau C, Osdoit M, van der Noordaa M, Shad S, Wei J, de Croze D, Hamy AS, Lae M, Reyal F, Sonke GS, Steenbruggen TG, van Seijen M, Wesseling J, Martin M, Del Monte-Millan M, Lopez-Tarruella S; I-SPY 2 Trial Consortium; Boughey JC, Goetz MP, Hoskin T, Gould R, Valero V, Edge SB, Abraham JE, Bartlett JMS, Caldas C, Dunn J, Earl H, Hayward L, Hiller L, Provenzano E, Sammut SJ, Thomas JS, Cameron D, Graham A, Hall P, Mackintosh L, Fan F, Godwin AK, Schwensen K, Sharma P, DeMichele AM, Cole K, Pusztai L, Kim MO, van 't Veer LJ, Esserman LJ, Symmans WF. Residual cancer burden after neoadjuvant chemotherapy and long-term survival outcomes in breast cancer: a multicentre pooled analysis of 5161 patients. Lancet Oncol. 2022 Jan;23(1):149-160. doi: 10.1016/S1470-2045(21)00589-1. Epub 2021 Dec 11. PMID 34902335
- [Background] Hudis CA, Barlow WE, Costantino JP, Gray RJ, Pritchard KI, Chapman JA, Sparano JA, Hunsberger S, Enos RA, Gelber RD, Zujewski JA. Proposal for standardized definitions for efficacy end points in adjuvant breast cancer trials: the STEEP system. J Clin Oncol. 2007 May 20;25(15):2127-32. doi: 10.1200/JCO.2006.10.3523. PMID 17513820
- [Background] Wolff AC, Somerfield MR, Dowsett M, Hammond MEH, Hayes DF, McShane LM, Saphner TJ, Spears PA, Allison KH. Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer. Arch Pathol Lab Med. 2023 Sep 1;147(9):993-1000. doi: 10.5858/arpa.2023-0950-SA. PMID 37303228